CLINICAL TRIAL: NCT06207760
Title: Targeting Inflammation in Depression Using Minocycline: a Patient Stratification Approach Using Peripheral Inflammatory Biomarkers, PET and MRI
Brief Title: Effect of Minocycline on Inflammation in Depressed Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Centro San Giovanni di Dio Fatebenefratelli (Other)
Collaborators: Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Annamaria Cattaneo, PhD, Lab head of Biological Psichiatry Unit, IRCCS Centro San Giovanni di Dio Fatebenefratelli
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RF-2018-12365308
Record Dates: First submitted 2023-11-27; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Minocycline

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Minocycline (Experimental): All subjects will receive Minocycline over 8 weeks in addition to their current antidepressant treatment.
  Interventions: Drug: Minocycline

INTERVENTIONS:
Drug: Minocycline — Minocycline (200 mg/day) for 8 weeks with a single daily administration (2 hard capsules of 100 mg)

SUMMARY:
The study aims to evaluate or to assess:

* An improvement in the peripheral inflammatory levels in depressed patients after 8 weeks of treatment with Minocycline in addition to their current antidepressant treatment;
* Any improvements in depressive symptoms after 8 weeks of treatment with Minocycline given as adjuvant to the current antidepressant treatment;
* Changes in the inflammatory status in the brain (in terms of microglia activation with 11C PK PET) after 8 weeks of treatment with Minocycline in addition to the current patient's treatment;
* Possible structural and functional brain changes evaluated by MRI after 8 weeks of treatment with Minocycline given as adjuvant to the current patient's treatment;
* Whether changes in MRI, in microglia activation, and peripheral inflammation correlate with the improvement in depressive symptoms.

In order to achieve these, a total of 60 patients, male and female, aged 25-45, who have not responded to their pharmacological treatment and who have medium-high levels of inflammation (with CRP> 2 mg/L) will be included in the study.

Enrolled patients will receive, in addition to their current antidepressant treatment, Minocycline (200 mg/day as total dosage) for 8 weeks.

Patients will be subjected to blood collection and clinical evaluations at baseline and after 8 weeks of treatment with Minocycline.

A subgroup of patients will be subjected to MRI and 11C PK PET assessment at baseline and after 8 weeks of treatment with Minocycline.

ELIGIBILITY:
Inclusion Criteria:

1. Being male or female depressed patients (aged 25-45);
2. Having a current DSM-V diagnosis of non-psychotic major depressive disorder confirmed by SCID;
3. Being non-responder to a current SSRI for at least 8 weeks, and historically to one other SSRI;
4. Being in stable antidepressant therapy for at least 8 weeks;
5. Being tolerant to the current SSRI;
6. Accepting Minocycline treatment;
7. Having CPR level> 2 mg/L;
8. Having signed and dated an informed consent to participate in the study;
9. Having no contraindications to receive treatment with Minocycline;
10. Having no contraindications to undergo the 11C-PK PET scan.

Exclusion Criteria:

1. Having active suicidal ideation;
2. Having a primary diagnosis of bipolar disorder, obsessive-compulsive disorder, eating disorder, PTSD;
3. Having a history of substance/alcohol abuse;
4. Having received tetracycline therapy within the previous 2 months;
5. Having a history of sensitivity to this class of drugs;
6. Having acute infections or an autoimmune or inflammatory disorder;
7. Having CRP>20 mg/L, as indicates acute infection or other major pathology;
8. Being sensitive to Minocycline;
9. Having a history of severe allergy or hypersensitivity to drugs;
10. Being hypersensitive to the active substance, to other tetracyclines or to any of the excipients;
11. Having severe renal failure;
12. Having hepatic dysfunction;
13. Being pregnant and in lactation;
14. (for MRI) Having pacemakers, electromechanical devices, ferromagnetic vascular clips, cochlear implants, stapedial prostheses, ferromagnetic foreign bodies, sickle cell anemia;

    EXCLUSION CRITERIA (FOR ONLY THOSE PATIENTS WHO WILL PERFORM 11C PK PET)
15. Having undergone imaging or treatment procedures using radiopharmaceuticals 7 days prior to the imaging session of this study;
16. Being unable to complete the 11C PK PET session, according to the clinician;
17. Being in current or previous (last two months) treatment with neuroactive drugs (benzodiazepines, barbiturates, picrotoxin and muscimol);
18. Being women of childbearing potential who are not surgically sterile and who do not guarantee to abstain from sexual activity for the 24 hours following the administration of 11C PK PET.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-28 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in the peripheral inflammatory status assessed by the measurement of CRP levels and inflammatory markers (i.e. IL-1, IL-6, IL-17 and TNF-alpha) | Changes from baseline to week 8
  To evaluate an improvement in the peripheral inflammatory status in depressed patients after 8 weeks of treatment with Minocycline in addition to their current pharmacological treatment.

SECONDARY OUTCOMES:
Change from baseline in depressive symptoms assessed by HAM-D17 | Changes from baseline to week 8
  To assess any improvements in depressive symptoms after 8 weeks of treatment with Minocycline given as adjuvant to the current antidepressant treatment.
Changes from baseline in central inflammatory levels by PET and by assessing differences in PK11195 binding | Changes from baseline to week 8
  To evaluate changes in the inflammatory status in the brain (in terms of microglia activation with 11C PK PET) after 8 weeks of treatment with Minocycline in addition to the current patient's treatment;
Structural and functional brain changes by MRI | Changes from baseline to week 8
  To evaluate by MRI possible structural and functional brain changes after 8 weeks of treatment with Minocycline given as adjuvant to the current patient's treatment.
Changes from baseline of the associations among brain structure observed with MRI, activation of microglia by PET, peripheral inflammatory markers and depression assessment scales | Changes from baseline to week 8
  Identification of correlations between a reduction of peripheral inflammation (by CRP and cytokines levels in blood samples) and/or central inflammatory status (by MRI and PET) and an improvement in depressive symptoms (evaluated by HAM-D17, SCID-5, BDI-II, STAI and CGI scale), after 8 weeks of treatment with Minocycline. Correlations will be calculated by using Pearson or Spearman correlation coefficients (statistical measures to analyse the relationship between variables with different units of measurement).

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Centro San Giovanni di Dio Fatebenefratelli, Brescia, Italy

IPD SHARING:
Plan to Share IPD: Undecided